CLINICAL TRIAL: NCT04310072
Title: Effects of Neuromuscular Electrostimulation in Patients With Acute Heart Failure - Results of a Single-centre Randomized Trial
Brief Title: Effects of Neuromuscular Electrostimulation in Patients With Acute Heart Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ploesteanu Rodica Lucia (Other)
Responsible Party: Sponsor-Investigator, Ploesteanu Rodica Lucia, principal investigator, Sfantul Pantelimon Emergency Hospital
Organization: Sfantul Pantelimon Emergency Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: SfantulPantelimon
Record Dates: First submitted 2020-03-09; First posted 2020-03-17 (Actual); Last update posted 2020-03-18 (Actual); Status verified 2020-03

CONDITIONS: Heart Failure
Keywords: Cardiac rehabilitation; Nouromuscular electrical stimulation
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Intervention Model Description: The study team conducted a prospective randomized study to investigate the effects of NMES versus standard therapy on a hospitalized population with AHF. After the patients with AHF were stabilized they were included in the trial and were randomized by a blinded investigator to control group or NMES therapy. At the time of enrollment, patients were clinically evaluated and their associated comorbidities and drug therapy were noted. ECG, echocardiography, 6-minute walk test (6MWT) were performed and laboratory samples were collected including oxidized LDL, NT- proBNP, CK, uric acid, lipid profile and PCR. At the time of discharge, all patients underwent a 6MWT and laboratory samples such as oxidized LDL and NT-proBNP were collected again. During the hospitalization period we monitored any adverse events and tolerance to NMES therapy. At the time of inclusion in the study, patients signed an informed consent form in two copies, one remaining with the patient.
Who Masked: Outcomes Assessor
Masking Description: After the patients were evaluated for inclusion in the study and after signing the informed consent form, they were randomized using the website www.randomization.com (1 complete randomized block). Considering our intervention protocol, it was not possible to blind the patients and/or the investigator who performed the electrostimulation. However, the other investigators who conducted the 6MWT and performed the randomization were blinded.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- neuromuscular electrical stimulation group (Experimental): For patients who underwent NMES therapy, four electrodes (two 50/100 mm and two 50/50 mm, Compex Performance) were placed on the skin above the quadriceps muscle approximately 5 cm below the inguinal fold and 3 cm above the upper patella border.
  The electrical stimulation protocol consisted of electrical current at frequency of 10 Hz, 20 seconds stimulation time (time on) and 20 seconds resting time (time off) with variable intensity (until visible muscular contraction) for one hour per day until discharge (Compex).The NMES therapy was on top of conventional rehabilitation described below.
  Interventions: Device: Neuromuscular electrical stimulation
- Control group (No Intervention): The control group consisted of patients who performed daily active upper and lower limbs exercise in bed and in a stand position (3x10 repetitions, "somewhat hard" on the Borg scale).

INTERVENTIONS:
Device: Neuromuscular electrical stimulation — NMES therapy induces visible rhythmic and repeated muscle contractions without volitional effort from the patient by applying electrodes to the thigh and/or calf muscles.
  Arms: neuromuscular electrical stimulation group

SUMMARY:
The investigators evaluated the effects of neuromuscular electrical stimulation (NMES) therapy on functional capacity and oxidative stress in patients hospitalized for an episode of acute heart failure (AHF). The NMES therapy was used on top of the conventional rehabilitation program. After randomization the investigators followed the patients by measuring the evolution of functional capacity, oxidative stress and adverse events.

DETAILED DESCRIPTION:
In this program the investigators will include patients with acute heart failure (AHF) with left ventricular ejection fraction (LVEF) lower than 50%, admitted to our clinic.

Patients prior to being included in this research will sign an informed consent form in two samples, one remaining with the patient. This form will contain the study protocol, risks, potential benefits as well as assuring patients that personal data will be used strictly for research purposes. The inclusion and exclusion criteria are presented below. The patients will be randomized into two groups: neuromuscular electrostimulation (NMES) therapy and conventional rehabilitation or a conventional rehabilitation program alone (respiratory gymnastics and strength / endurance exercises in bed).

Patients will receive optimal medical therapy for AHF according to current management guidelines. Patients will complete different questionnaires (Kansas, Beck for Depression). In the first phase, patients will be given a form with questions regarding notions about heart failure and cardiovascular recovery to assess the level of knowledge about their disease.

All patients included will perform the following:

* Clinical evaluation
* ECG
* Biological samples (including NT pro BNP, CK, oxidized LDL plus standard samples)
* Cardiac ultrasound
* 6-minute walk test (6MWT) The duration of NMES therapy will be equal to the duration of hospitalization. At the time of discharge, all patients will undergo a 6MWT and biological samples (NT pro BNP and oxidized LDL) and receive a cardiac rehabilitation program that they will follow at home. They will be given advice on initiating and maintaining a healthy diet, as well as discontinuing smoking if this risk factor is identified.

There will be a telephone visit at 30 days and the investigator will note the vital status and rehospitalizations.

ELIGIBILITY:
Inclusion Criteria:

* patients with acute heart failure and a LVEF below 50% (echocardiography), admitted consecutively to the cardiology clinic of "Sfantul Pantelimon" Hospital, Bucharest

Exclusion Criteria:

* age under 18 years,
* acute coronary syndrome in the last month,
* recent myocardial revascularization (in the last 6 weeks),
* severe ischemic lesions at the level of the lower limbs,
* life-threatening arrhythmias,
* uncontrolled blood pressure,
* high-grade atrioventricular block,
* acute myocarditis,
* acute pericarditis,
* obstructive hypertrophic cardiomyopathy,
* acute systemic disease,
* deep vein thrombosis,
* severe uncorrected primary valvular disease,
* psychiatric disorders or marked cognitive impairment,
* active neoplastic disorders except basal or squamous cell carcinoma,
* other conditions that in the opinion of the investigator do not allow the participation to the study
* patient's refusal.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-09-10 (Actual); Primary Completion 2019-11-20 (Actual); Study Completion 2019-11-20 (Actual)

PRIMARY OUTCOMES:
evaluate the impact of NMES therapy applied during hospitalization on the functional capacity | up to one month (30 days)
  The investigators will measure 6 minute walk test at the inclusion in the trial ans at the time of discharge
evaluate the impact of NMES therapy on oxidative stress | up to one month (30 days)
  The investigator will measure oxidized LDL plasmatic levels at the inclusion in the trial ans at the time of discharge

CONTACTS AND LOCATIONS:
Overall Officials: Mihai Berteanu, Principal Investigator — Elias Emergency Hospital
Locations (1):
- Spitalul Sfantul Pantelimon, Bucharest, București, Romania

IPD SHARING:
Plan to Share IPD: Yes
All the individual participant data can be available by email on request. This study is a part of a PhD thesis and a publication of the results will follow
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The data is available from the present and 15 years from now
Access Criteria: all the data can be accessed by request on email

REFERENCES:
- [Result] Ploesteanu RL, Nechita AC, Turcu D, Manolescu BN, Stamate SC, Berteanu M. Effects of neuromuscular electrical stimulation in patients with heart failure - review. J Med Life. 2018 Apr-Jun;11(2):107-118. PMID 30140316